CLINICAL TRIAL: NCT05442892
Title: Use of Near Infrared Spectroscopy (NIRS) as a Biomarker of Delirium in Hospitalized Older Adults Applied to a Multicomponent Program Based on Physical Exercise
Brief Title: Use of Near Infrared Spectroscopy (NIRS) as a Biomarker of Delirium in Hospitalized Older Adults Doing Physical Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Miguel Servet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DelNIRS
Record Dates: First submitted 2022-06-14; First posted 2022-07-05 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Delirium
Keywords: physical exercise; multicomponent intervention; geriatric acute unit; older adults
MeSH Terms: conditions — Delirium; Motor Activity

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physical exercise (Experimental): The intervention will consist of a multicomponent exercise training programme, which will be composed of supervised progressive resistance exercise training, balance-training, strength-training and walking for 4 consecutive days. During the training period, patients will be trained in 30 min sessions daily.
  Interventions: Procedure: Multicomponent exercise training programme
- Without physical exercise (No Intervention): Participants randomly assigned to the usual care group will receive normal hospital care, which includes physical rehabilitation when needed

INTERVENTIONS:
Procedure: Multicomponent exercise training programme — The supervised multicomponent exercise training programme will be comprised of upper and lower body strengthening exercises, tailored to the individuals functional capacity, using weight machines and aiming for 2-3 sets of 8-10 repetitions at an intensity of 30-60% of 1RM (Matrix, Johnson Health Tech, Ibérica, S.L. Torrejón de Arroz, Madrid, Spain) combined with balance and gait retraining exercises that progressed in difficulty and functional exercises such as rises from a chair.
  Arms: Physical exercise

SUMMARY:
Delirium is an important cause of morbimortality in older adults admitted to hospital. Multicomponent interventions targeting delirium risk factors, including physical exercise and mobilization, have been shown to reduce delirium incidence in 30-40% in acute care setting but little is known about its role in the evolution of delirium, once established.

This study is a randomized clinical trial conducted in the Acute Geriatric Unit of a tertiary public hospital in Navarra, Spain. Hospitalized delirious patients who meet the inclusion criteria will be randomly assigned to the intervention or control group. The intervention will consist of a multicomponent exercise training programme, which will be composed of supervised progressive resistance and strength exercise training during 4 consecutive days. The objective is to assess the effectiveness of this intervention in reducing the following primary outcomes: duration and severity of delirium, functional status, and length of stay.

This study will contribute to determine the usefulness of physical exercise in the management of delirium. It will be the first study to evaluate the impact of a multicomponent intervention based on physical exercise in the evolution of delirium.

DETAILED DESCRIPTION:
This study is a randomized clinical trial conducted in the Acute Geriatric Unit of Navarra University Hospital (Pamplona, Spain) with 40 beds allocated. Hospitalized patients who meet the inclusion criteria will be randomly assigned to the intervention or control group. After signing an informed consent form, the participants will be randomly assigned to either the intervention or control group. The data for both the intervention and the control group will be obtained at five different times: the initial visit during the acute hospitalization, at discharge and at one, three and twelve months after discharge through phone call and clinical history. Adverse events, including muscle pain, fatigue, falls and general aches will be recorded by the training staff.

Delirium will be assessed using the European Spanish version of the 4AT daily during hospitalization until discharge. This tool has been validated for the Spanish population and is a reliable instrument for delirium detection in older patients. Delirium severity will be evaluated with the Memorial Delirium Assessment Scale (MDAS) which is also validated in Spain.

Therefore, brain function will be examinated during delirium and the effects of an intra-hospital exercise program on the prefrontal cortex region and also on muscle function with the use of functional near-infrared spectroscopy imaging (NIRS). Regional cerebral oxygen saturation (Scto2) will be recorded using NIRS through the NIRO-200NX C10448 monitor (Hamamatsu, Japan) by placing one optode on the patient's forehead above the eyebrow (contralateral to the dominant hand) and the other optode on the vastus lateralis muscle. The measurements will be made with the patients resting in the sitting position after 60 seconds, doing trail making test part A and physical exercise at the beginning of the study and at the 4th day of the study, in both intervention and control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 75 years admitted to the Geriatric Service of the Navarra University Hospital for at least 4 days

Exclusion Criteria:

* Refusal to sign the informed consent by the patient/primary caregiver/legal representative or inability to obtain it
* Advanced dementia GDS 6-7
* Moderate functional impairment (Barthel Index less than 45)
* Life expectancy less than 3 months
* Facial dermal pathology
* Acute intracranial pathology (hemorrhages, cerebral infarcts)
* Recent acute myocardial infarction
* Unstable angina
* Severe heart valve insufficiency
* Arrhythmia or uncontrolled arterial hypertension
* Recent pulmonary thromboembolism
* Hemodynamic instability

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Changes in the 4 'A's Test (4AT scale Spanish version) | 12 months
  The change in the 4 'A's Test (4AT scale) measured at baseline and follow-up. The 4AT is designed to be used as a delirium detection tool in general clinical settings.The 4AT has 4 parameters: Alertness, Abbreviated mental test-4 (AMT4), Attention (months backwards test) and Acute change or fluctuating course. The score range is 0-12, with scores of 4 or more suggesting possible delirium. Scores of 1-3 suggest possible cognitive impairment.
Changes in the Memorial Delirium Assessment Scale (MDAS scale Spanish version). | 12 months
  The change in Memorial Delirium Assessment Scale (MDAS scale Spanish version) measured at baseline and follow-up. MDAS scale was designed to diagnose delirium as well as classify delirium severity. The instrument reflects delirium diagnostic criteria from DSM. It has 10 severity items rated 0 to 3 points for a maximum total score of 30 points, with higher scores representing more severe delirium.

SECONDARY OUTCOMES:
Change in functional capacity: Barthel Index (Spanish version) | 12 months
  The change in Barthel Index measured at baseline and follow-up (a measure of Basic Activities of Daily Living). This index ranges from 0 worst to 100 best.
Change in cognitive status: Informant Questionnaire on Cognitive Decline in the Elderly-short form (IQCODE-short form Spanish version) | 12 months
  The change in IQCODE-short form will be measured at baseline and follow-up. This test has 16 questions. Each question is scored from 1 (much improved) to 5 (much worse). For the Short IQCODE, a cut-off point (average score) of 3.31/3.38 achieves a balance of sensitivity and specificity of cognitive impairment.
Change in quality of life measured by the Spanish version of the EuroQol-5 Dimension (EQ-5D) questionnaire | 12 months
  The change in EuroQol-5 Dimension (EQ-5D) questionnaire measured at baseline and follow-up. The EQ records the respondent´s overall current health on a vertical visual analogue scale, where the endpoints are labelled "The best health you can imagine" and "The worst health you can imagine". Minimum 0 Maximum 100 Higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Lozano Vicario, MD, Principal Investigator — Hospital Universitario de Navarra (Pamplona, Spain)
Locations (1):
- Hospital Universitario de Navarra (HUN), Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in delirium and frailty. Data or samples shared will be coded.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).

REFERENCES:
- [Derived] Lozano-Vicario L, Zambom-Ferraresi F, Zambom-Ferraresi F, de la Casa-Marin A, Ollo-Martinez I, Saez de Asteasu ML, Cedeno-Veloz BA, Fernandez-Irigoyen J, Santamaria E, Romero-Ortuno R, Izquierdo M, Martinez-Velilla N. Effectiveness of a multicomponent exercise training program for the management of delirium in hospitalized older adults using near-infrared spectroscopy as a biomarker of brain perfusion: Study protocol for a randomized controlled trial. Front Aging Neurosci. 2022 Dec 15;14:1013631. doi: 10.3389/fnagi.2022.1013631. eCollection 2022. PMID 36589545